CLINICAL TRIAL: NCT02687165
Title: Uncovering Neural and Immune Mechanisms of Chronic Pain in Post Treatment Lyme Syndrome
Acronym: PTLS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment due to strict inclusion/exclusion criteria
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Alla Landa, Assistant Professor, New York State Psychiatric Institute
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 7003; NCT05055622 (obsolete NCT alias)
Record Dates: First submitted 2016-02-16; First posted 2016-02-22 (Estimated); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Post Treatment Lyme Syndrome (PTLS); Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Milnacipran; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milnacipran augmented by D-cycloserine (Active Comparator): participants will be receiving Milnacipran for 12 weeks. During weeks 6-12 participants will be receiving D-cycloserine in addition to Milnacipran
  Interventions: Drug: Milnacipran and D-cycloserine
- Milnacipran augmented by Placebo (Placebo Comparator): participants will be receiving Milnacipran for 12 weeks. During weeks 6-12 participants will be receiving placebo in addition to Milnacipran
  Interventions: Drug: Milnacipran and D-cycloserine

INTERVENTIONS:
Drug: Milnacipran and D-cycloserine — Milnacipran augmented by D-cycloserine

SUMMARY:
This study will investigate (a) neural and immune mechanisms underlying chronic pain in PTLS by comparing a group of PTLS patients and healthy participants on brain imaging, sensory, and immune markers; and (b) assess change in pain, brain imaging (fMRI and MRS), sensory, and immune markers in response to a combination of SNRI and glutamatergic treatment for chronic pain in PTLS (Milnacipran and D-cycloserine).

DETAILED DESCRIPTION:
At least 5-15% of patients with Lyme disease (7,500-45,000 new cases a year) develop Post-treatment Lyme Syndrome (PTLS) - debilitating residual symptoms that last months to years, even after having received antibiotic treatment. Often patients with PTLS experience chronic pain in their muscles or joints or nerves.

Because many PTLS patients have pain that persists despite antibiotics and because we know that medicines which modulate the pain pathways in the brain can help to reduce or eliminate pain, we plan to treat patients with a medicine that is FDA approved for the treatment of pain. This medicine is known as Milnacipran (the trade name is "Savella"); this medicine is not addictive and it has been shown to reduce chronic pain by its multiple actions on pain pathways. All patients in the study will be treated with this FDA approved medicine.

Second, we wish to test whether the pain can be improved even further by adding a medicine which is known to modulate the glutamate transmission involved with pain in the brain. This medicine - D-Cycloserine - is actually an antibiotic, currently FDA approved for the treatment of tuberculosis. Because of its action on glutamate receptors, we are hypothesizing that it will help to decrease pain even further in patients with Lyme-related pain. In order to test this hypothesis, after 6 weeks of being on Milnacipran, all patients will then be given an additional treatment - either D-Cycloserine or a placebo pill (a placebo is a pill that does not contain any active medication.) At the end of 12 weeks, we will then evaluate improvement compared to when the patient started in the study using the same clinical and neuroimaging (fMRI) tests.

Finally, we want to know whether patients with PTLS have over-active central pain circuits in the brain. Because pain is processed through the brain's pain circuits, we wish to examine whether people suffering from PTLS have hyper-active pain circuits that make them more sensitive to pain than those who have normally-active pain circuits. To do this, we will be comparing patients with PTLS to healthy volunteers by conducting careful neurologic and brain imaging (fMRI) studies.

We hope that this study will provide valuable information about how the brain processes pain signals in PTLS and about whether this treatment approach is effective.

ELIGIBILITY:
Inclusion Criteria:

1. History of Lyme Disease and treatment:
2. Current chronic pain in the musculoskeletal system
3. clinically troubling sensory hypersensitivity (e.g., light or touch)
4. Able to speak and read English
5. Willing to not take other than study centrally acting pharmacologic agents prior to MRI and for the duration of treatment with study medications

Exclusion Criteria:

1. Diagnosis of another (not LYME) general medical condition that has a major role in the onset, severity, exacerbation or maintenance of pain, or sensory hypersensitivity.
2. DSM-IV Axis I lifetime diagnosis of Pervasive Developmental Disorder, Autism, Psychotic disorder, Bipolar Disorder, Substance dependence.
3. I current diagnosis of Major Depressive Disorder or substance abuse
4. History of head injury with loss of consciousness (>5min), neurologic disease, seizures (excluding febrile seizures) or serious unstable medical condition (e.g. cancer, diabetes)
5. Current or recent (last month) opiate use
6. For 2 weeks prior to MRI and diagnostic visit, unable to be free of centrally active medications or treatment methods. These include medications commonly used to treat pain (eg, antidepressants, muscle relaxants, centrallyacting analgesics), as well as transcutaneous electrical nerve stimulation, biofeedback, tender and trigger point injections, acupuncture, and anesthetic or narcotic patches. PRN doses of short acting medications, e.g. acetaminophen, aspirin, and nonsteroidal antiinflammatory agents will be allowed for pain with usage carefully monitored, but patients must be willing to be off of these medications for 24 hours prior to the major evaluations at intake and MRI study visit. Stable doses of non-benzodiazepines will be allowed for sleep (but not tricyclics)
7. Ferromagnetic implants (e.g. pacemaker, etc.)
8. Metal Braces or Retainers
9. Transdermal medicinal patches that cannot be removed
10. Birth at < 37 weeks gestational age (prior studies have shown dramatic effects on brain structure and function in prematurely born children)
11. Claustrophobia
12. Women will be excluded if they are pregnant, lactating, or not either surgically-sterile or using appropriate methods of birth control. Women must agree to continue using applicable birth control throughout the trial. All women of child-bearing potential must have a negative pregnancy test at the intake visit.
13. Inability to reliably rate intensity of pain in response to a fixed thermal stimulus
14. Inability to tolerate sound intensity of fMRI
15. Individuals currently successfully treated by medications for their pain.
16. History of inability to tolerate treatment with SSRI or SNRI medications or d-cycloserine; or medication induced mania
17. Renal insufficiency or congestive heart failure
18. Hepatic malfunction Liver Test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 patients were screened, but none was randomized
Pre-assignment Details: 4 patients were screened, but no one was randomized
Period: Overall Study
Arm/Group | Milnacipran Augmented by D-cycloserine | Milnacipran Augmented by Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No one was randomized.
Groups:
- All Participants: participants were not randomized. reporting all subjects together.
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Data were not collected
  Participants
    Female | 2
    Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory
Description: average pain over past week on the scale from 0-10. Data were not collected.
Time Frame: 12 weeks
Population: patients didn't compete the study. Data were not collected.
Arm/Group | Milnacipran Augmented by D-cycloserine | Milnacipran Augmented by Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Only some baseline demographic information were collected. And no subject was randomized. Study terminated.
Description: Adverse events were not monitored/assessed. 0 Participants at Risk.
Arm/Group | Milnacipran Augmented by D-cycloserine | Milnacipran Augmented by Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No